CLINICAL TRIAL: NCT02277899
Title: Primary Care, Communication, and Improving Children's Health
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1K23HL118152-01A1 Aim 2; 1K23HL118152-01A1 (NIH)
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Childhood Obesity; Overweight; Communication; Weight Loss
Keywords: childhood obesity; overweight; communication; primary care; weight management; communication methods; patient-centered communication
MeSH Terms: conditions — Pediatric Obesity; Overweight; Communication; Weight Loss | interventions — Counseling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Overweight school-age children: Overweight 6-12 year-old children. Weight status will be measured and parents complete surveys at baseline and one year later. Pediatricians will complete surveys at baseline, and after index visit. Visits will be directly video-recorded.
  The impact of pediatrician clinical practices and communication strategies on child's weight status will be evaluated at one year. Clinical practices (such as risk-factor screening) that occur during the 1-year interval between well-child visits also will be assessed. Specific clinical practice elements and communication strategies that will be examined include:
  1. Communication regarding child's high weight status
  2. Counseling regarding cardiovascular risk factor screening and assessment
  3. Behavioral counseling
  4. Interval follow-up to readdress weight, and
  5. Patient-centeredness, scored as the ratio of patient to doctor-centered communication regarding weight topics.
  Interventions: Other: Communication regarding overweight status; Other: Risk-factor assessment and counseling; Other: Lifestyle behavior assessment and counseling; Other: Interval follow-up to readdress weight; Other: Patient-centered communication

INTERVENTIONS:
Other: Communication regarding overweight status — Pediatrician-patient/parent communication regarding child's high weight status
Other: Risk-factor assessment and counseling — Counseling regarding cardiovascular risk factor assessments/results.
Other: Lifestyle behavior assessment and counseling — Counseling regarding diet and lifestyle changes to improve weight status.
Other: Interval follow-up to readdress weight — Interval follow-up to readdress weight, prior to the next well-child visit one year later. Follow-up could include ongoing care through nutrition and/or an intensive weight-management program.
Other: Patient-centered communication — Patient-centered communication will be scored as the ratio of patient to doctor-centered communication regarding weight topics. Means will be calculated for total and weight-communication-specific pediatrician, child, and parent-talk time, and patient, doctor, and the ratio of patient/doctor-centered communication scores. For the primary hypothesis, biomedical information-giving (for example, risk-factor communication) will be treated as patient-centered because the principal investigator's focus groups suggest that parents want this information, and prior research suggests that including biomedical-information giving improves the correlation of Roter's patient-centeredness measure with patient health status and satisfaction scores.

SUMMARY:
The purpose of this study is to determine communication content and strategies in primary care that predict improvement in weight status among overweight school-age children.

DETAILED DESCRIPTION:
We will test whether 1) pediatrician-patient communication regarding overweight status, behavior/risk-factor counseling, and the frequency and time to next follow-up visit, compared with either no communication or incomplete communication (communicating only high weight status without behavior/risk-factor counseling or a follow-up visit) will predict improvement in weight status at one year follow-up, and 2) during pediatrician-patient communication regarding weight and weight management, higher patient-centeredness will predict improvement in weight status at one year follow-up. The communication content identified will generate new information about the most effective content and style of pediatrician-patient communication that predict weight-status improvement. Because we prospectively will examine clinical practice elements in the one-year interval between well-child visits, acknowledging that communication regarding high weight status may initiate assessment of risk factors for heart disease (such as high cholesterol and blood sugar), more frequent follow-up visits, or prompt a nutrition referral, we will generate novel information about the most effective clinical practices and follow-up interval and frequency that predict weight-status improvement in overweight children. We also will examine if the content and style of communication are related to improvements in diet and lifestyle behaviors at one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Schedule a well-child visit with a participating pediatrician
* Agree to return in one year for the follow-up well-child visit
* Overweight
* 6-12 years old
* Have a working telephone and/or e-mail address
* Child/parent willing to provide assent/consent

Exclusion Criteria:

* Unstable illness (such as uncontrolled asthma)
* Developmental condition (such as trisomy 21)
* Planning to move/leave practice within two years

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We will recruit pediatricians (from academic, community, and private practices), children, and a consenting parent. Pediatricians and children will be selected to reflect the proportions of minority pediatricians and children in the practices. Pediatricians at the community and private practices will be eligible to participate if they provide outpatient pediatric care ≥20 hours/week. At the academic clinic, only second and third-year residents will be eligible. Eighty-five children and a consenting parent will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Percent overweight | From recorded well-child visit to next well-child visit, approximately 12 months later
  The percent over the median BMI percentile for age and gender. This measure changes comparably for similar weight changes in overweight and severely-obese children. In contrast, an overweight child would have to lose substantially less weight than a severely-obese child for the same change in BMI z-score.

SECONDARY OUTCOMES:
BMI z-score | From recorded well-child visit to next well-child visit, approximately 12 months later
  Change in BMI z-score of 0.25-0.5 has been associated with reductions in cardiovascular-disease risk factors. Using both percent overweight and BMI z-score measures will allow examination of the relationship between relative weight changes and cardiovascular-disease risk-factor improvement.

OTHER OUTCOMES:
Change in the number of "5-2-1-0" behaviors | From recorded well-child visit to next well-child visit, approximately 12 months later
  The "5-2-1-0" behaviors are: eat five fruits and vegetables, watch "screens" (TV, computer, tablets, video games, cell phones, etc…) two hours per day or less, be physically active for one hour per day or more, and drink zero calorie-containing beverages per day.

CONTACTS AND LOCATIONS:
Overall Officials: Christy B Turer, MD, MHS, Principal Investigator — University of Texas Southwestern and Children's Medical Center Dallas
Locations (1):
- University of Texas Southwestern and Children's Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Turer CB, Montano S, Lin H, Hoang K, Flores G. Pediatricians' communication about weight with overweight Latino children and their parents. Pediatrics. 2014 Nov;134(5):892-9. doi: 10.1542/peds.2014-1282. Epub 2014 Oct 13. PMID 25311599
- [Background] Turer CB, Mehta M, Durante R, Wazni F, Flores G. Parental perspectives regarding primary-care weight-management strategies for school-age children. Matern Child Nutr. 2016 Apr;12(2):326-38. doi: 10.1111/mcn.12131. Epub 2014 Apr 10. PMID 24720565
- [Background] Upperman C, Palmieri P, Lin H, Flores G, Turer CB. What do parents want for their children who are overweight when visiting the paediatrician? Obes Sci Pract. 2015 Oct;1(1):33-40. doi: 10.1002/osp4.5. Epub 2015 Sep 10. PMID 28580163
- [Background] Turer CB, Upperman C, Merchant Z, Montano S, Flores G. Primary-Care Weight-Management Strategies: Parental Priorities and Preferences. Acad Pediatr. 2016 Apr;16(3):260-6. doi: 10.1016/j.acap.2015.09.001. Epub 2015 Sep 26. PMID 26514648
- [Background] Turer CB, Barlow SE, Montano S, Flores G. Discrepancies in Communication Versus Documentation of Weight-Management Benchmarks: Analysis of Recorded Visits With Latino Children and Associated Health-Record Documentation. Glob Pediatr Health. 2017 Feb 6;4:2333794X16685190. doi: 10.1177/2333794X16685190. eCollection 2017. PMID 28239625